CLINICAL TRIAL: NCT02212405
Title: Does the Insula Control Smoking-Induced Dopamine Release? A TMS/[11C]-PHNO Study in Humans (Part II).
Brief Title: Does the Insula Control Smoking-Induced Dopamine Release? A TMS/[11C]-PHNO Study in Humans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Brainsway (Industry)
Responsible Party: Principal Investigator, Bernard Le Foll, Principal investigator, MD, PhD, CCFP, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 170/2010
Record Dates: First submitted 2014-07-30; First posted 2014-08-08 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Deep rTMS; Insular cortex; PET; [11C]-PHNO
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- rTMS Sham + PET (Sham Comparator): An advanced sham coil will be used that mimicks the sound and sensation of real repetitive Transcranial Magnetic Stimulation. The repetitive Transcranial Magnetic Stimulation sham intervention is followed by radiotracer and PET.
  Interventions: Other: repetitive Transcranial Magnetic Stimulation Sham
- rTMS 1Hz + PET (Experimental): Deep repetitive Transcranial Magnetic Stimulation will be applied to the insula for 30 minutes. This will consist of 20 trains each comprising of 50 pulses at 1Hz. The inter-train interval is 15 seconds. The intervention is followed by radiotracer and PET.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- rTMS 10Hz + PET. (Experimental): Deep repetitive Transcranial Magnetic Stimulation will be applied to the insula for 30 minutes. This will consist of 34 trains each comprising of 30 pulses at 10Hz. The inter-train interval is 3 seconds. The intervention is followed by radiotracer and PET.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — Each participant will participate in all three arms to receive sham, 1hz and 10hz rTMS as well as PET imaging.
  Other Names: Deep Repetitive Transcranial Magnetic Stimulation; DTMS HLRIADD-COIL, Model 102B
  Arms: rTMS 10Hz + PET.; rTMS 1Hz + PET
Other: repetitive Transcranial Magnetic Stimulation Sham — The sham coil is built in the same helmet of the active coil. The sham coil is has a circular shape and placed perpendicular to the scalp within the same helmet. This coil produces a similar sound and scalp sensation as the real coil.
  Arms: rTMS Sham + PET

SUMMARY:
Findings from this study may demonstrate how the insula contributes to reward pathways involved in addiction. There are three main hypotheses for this trial. The first is that inhibiting the insula using transcranial magnetic stimulation (TMS) will not cause noticeable changes of dopamine release in the striatum. The second is that stimulating the insula with TMS will increase dopamine release in the striatum, and will be visualized on PET imaging as decreased radiotracer binding. The third hypothesis is that the participants will not experience major side effects from TMS on the insula.

DETAILED DESCRIPTION:
This project will take advantage of the recently developed Deep rTMS coil to target the insular cortex. Few studies have examined the possibility of using repetitive Transcranial Magnetic Stimulation (rTMS) for nicotine addiction and none so far have explored the use of a coil that specifically targets the insular region. The objective of this study is to test whether low and high-frequency rTMS of the insula modulates striatal dopamine (DA) release in healthy humans. Positron Emission Tomography (PET) with [11C]-(+)-PHNO, a radiotracer which is very sensitive to fluctuations in DA transmission in the human brain, will be used to assess the impact of rTMS on dopamine levels. This project will yield the first data in humans linking the insula to the DA system in vivo. These findings could lead to the identification of optimal parameters for Deep rTMS to use secondarily in a proof of principle clinical study in smokers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Between the ages of 19 and 45

Exclusion Criteria:

* Pregnancy.
* Presence of metal objects in the body or implanted electronic devices, that preclude safe MR scanning.
* Claustrophobia.
* Cardiovascular or cerebrovascular diseases.
* Major psychiatric disorders including mood, anxiety or psychotic disorders.
* History of or current neurological illnesses including seizure disorders, migraine, multiple sclerosis, movement disorders, head trauma, CVA or CNS tumor.
* Gross structural brain abnormalities as revealed by T1 weighted images.
* Current use or use during the previous month of medication that may affect the CNS (e.g. neuroleptics, bupropion).
* Learning disability, amnesia or other conditions that impede memory and attention.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in [11C]-(+)-PHNO binding | Participants will complete all sessions in a period of approximately 4 weeks.
  [11C]-(+)-PHNO binding at D2/3 receptors will be measured with PET imaging following rTMS at 1Hz, 10Hz, and sham stimulation. Binding at regions of interest will be compared between trial conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard LeFoll, M.D., Ph.D, Principal Investigator — CAMH
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Malik S, Jacobs M, Cho SS, Boileau I, Blumberger D, Heilig M, Wilson A, Daskalakis ZJ, Strafella AP, Zangen A, Le Foll B. Deep TMS of the insula using the H-coil modulates dopamine release: a crossover [11C] PHNO-PET pilot trial in healthy humans. Brain Imaging Behav. 2018 Oct;12(5):1306-1317. doi: 10.1007/s11682-017-9800-1. PMID 29170944
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching — http://www.camh.ca/en/research/Pages/research.aspx